CLINICAL TRIAL: NCT00331695
Title: Evaluation of the Efficacy of 17 Alpha-hydroxyprogesterones Caproate for the Prevention of Preterm Delivery
Brief Title: Efficacy of 17 Alpha-hydroxyprogesterones Caproate for the Prevention of Preterm Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe AUCAN, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040438
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2007-03

CONDITIONS: Preterm Delivery
Keywords: Progesterone; Preterm delivery; Preterm labor; Cervical length; ultrasonography
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 17 alpha-hydroxyprogesterones caproate
  Interventions: Drug: 17 alpha-hydroxyprogesterones caproate

INTERVENTIONS:
Drug: 17 alpha-hydroxyprogesterones caproate — 17 alpha-hydroxyprogesterones caproate

SUMMARY:
To demonstrate that the intramuscular administration of 17 alpha hydroxyprogesterones caproate allows to reduce the risk of preterm delivery, in 3 high risk populations defined by the association of an ultrasonographic cervical length egal and inferiority 26 mm between 20 and 32 weeks of gestation and:

* either a first episode of preterm labor stopped by acute tocolysis;
* either a history of late miscarriage or premature delivery or uterine malformation or DES
* either a twin pregnancy. Therefore, a randomised, multicentre trial has been designed with initial stratification according to these three risk groups, opened with two parallel arms.

DETAILED DESCRIPTION:
Objective

To demonstrate that the intramuscular administration of 17 alpha - hydroxyprogesterones caproate allows to reduce the risk of preterm delivery, in 3 high risk populations defined by the association of an ultrasonographic cervical length 26 mm between 20 and 32 weeks of gestation and:

* either a first episode of preterm labor stopped by acute tocolysis;
* either a history of late miscarriage or premature delivery or uterine malformation or DES
* either a twin pregnancy. Experimental design Prospective, randomized, multicenter, trial with initial stratification according to three risk groups, opened with two parallel arms.

The maximal duration for treatment will be 16 weeks for each included patient. The duration for inclusions will be 30 months. The duration for participation of each patient will be 10 to 22 weeks. The foreseen inclusion period for this trial is from 06/01/2006 to 12/31/2008 Description Two therapeutic strategies will be compared in each risk group and attributed by uniform randomisation.

Arm A :IM injection of 17 alpha hydroxyprogesterones caproate, 500 mg, twice a week until 36 W or until preterm delivery in high risk symptomatic group and high risk twin pregnancies group.

IM injection of 17 alpha-hydroxyprogesterones caproate, 500 mg, once a week until 36 W or until preterm delivery in high risk asymptomatic group.

Arm B :No treatment with 17 alpha-hydroxyprogesterones caproate. (usual management) Presentation : Progesterone retard Pharlon 500 mg Tolerance criteria

* nausea,vomiting,
* weakness

ELIGIBILITY:
Inclusion Criteria:

* ultrasonographic cervical length 26 mm between 20 and 32 weeks of gestation and:
* either a first episode of preterm labor stopped by acute tocolysis
* either a history of late miscarriage or premature delivery or uterine malformation or DES;
* either a twin pregnancy.

Exclusion Criteria:

* cervical dilatation > 3 cm,
* chorioamnionitis,
* fetal distress,
* placenta praevia,
* abruptio placenta,
* preterm premature rupture of membranes,
* polyhydramnios,
* Twin-twin transfusion syndrome,
* IUGR,
* preeclampsia or hypertension,
* other pathology justifying a preterm delivery,
* epilepsy drugs
* participation to another therapeutic trial,
* any patient for whom informed consent cannot be obtained.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 560 (Actual)
Dates: Start 2006-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Interval between inclusion and delivery. | during de study
  Interval between inclusion and delivery.

SECONDARY OUTCOMES:
Preterm delivery rate < 37 W, < 34 W et < 32 W, | during the study
  Preterm delivery rate < 37 W, < 34 W et < 32 W,
Number of hospitalizations for preterm labor, | during the study
  Number of hospitalizations for preterm labor,
Cerclage performed at or after 20 weeks, | during the study
  Cerclage performed at or after 20 weeks,
Neonatal weight, | during the study
  Neonatal weight,
NICU transport | during the study
  NICU transport
Respiratory distress syndrome, | during the study
  Respiratory distress syndrome,
Bronchopulmonary dysplasia, | during the study
  Bronchopulmonary dysplasia,
Necrotizing enterocolitis, | during the study
  Necrotizing enterocolitis,
leucomalacia, | during the study
  leucomalacia,
neonatal death. | during the study
  neonatal death.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick ROZENBERG, MD,, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - CHI Poissy st Germain, Poissy
  - Chi Poissy St Germain, Poissy

REFERENCES:
- [Background] Rozenberg P, Rudant J, Chevret S, Boulogne AI, Ville Y. Repeat measurement of cervical length after successful tocolysis. Obstet Gynecol. 2004 Nov;104(5 Pt 1):995-9. doi: 10.1097/01.AOG.0000143254.27255.e9. PMID 15516390
- [Derived] Winer N, Bretelle F, Senat MV, Bohec C, Deruelle P, Perrotin F, Connan L, Vayssiere C, Langer B, Capelle M, Azimi S, Porcher R, Rozenberg P; Groupe de Recherche en Obstetrique et Gynecologie. 17 alpha-hydroxyprogesterone caproate does not prolong pregnancy or reduce the rate of preterm birth in women at high risk for preterm delivery and a short cervix: a randomized controlled trial. Am J Obstet Gynecol. 2015 Apr;212(4):485.e1-485.e10. doi: 10.1016/j.ajog.2014.10.1097. Epub 2014 Oct 30. PMID 25448515